CLINICAL TRIAL: NCT04967300
Title: Measuring and Evaluating the Changes in Anxiety Levels of Children With Repetitive Sessions of Dental Treatments: A Retrospective Observational Cohort Study
Brief Title: Measuring and Evaluating the Changes in Anxiety Levels of Children With Repetitive Sessions of Dental Treatments
Status: Completed | Type: Observational
Sponsor: Erzincan University (Other)
Responsible Party: Principal Investigator, Nurcan Kutluer Karaca, Assistant Professor Doctor, Erzincan University
Other Study IDs: Erzincan Binali Yıldırım U.
Record Dates: First submitted 2021-06-08; First posted 2021-07-19 (Actual); Last update posted 2021-07-19 (Actual); Status verified 2021-07

CONDITIONS: Dental Anxiety
MeSH Terms: interventions — Dental Care

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- First Visit: Children who visit dentist at first time
  Interventions: Procedure: Dental treatment
- Second Visit: Children who visit dentist at second time
  Interventions: Procedure: Dental treatment

INTERVENTIONS:
Procedure: Dental treatment — bilateral restorative treatment on the mandibular primary first molars

SUMMARY:
Dental anxiety is defined as the fear of terrible events during dental treatment and the loss of control.Anxiety may be related to adaptation of the patient to external factors in environment, so the adaptation of the pediatric patient to the stimuli in the dental environment may affect the level of anxiety.The aim of the this study was to evaluate the relationship between sequential visits in dental treatments and dental anxiety levels of pediatric patients with anxiety scales and physiological measurements.

DETAILED DESCRIPTION:
A total of 224 children aged 5-8 years who needed at least two restorative dental treatment of the mandibular first primary molar were included in the study.

In each sessions the Wong-Baker FACES Pain Rating Scale (W-BFRS) was used to evaluate the dental anxiety before and after the treatment.

The Modified Corah's Dental Anxiety Scale (MDAS) was used as a dental anxiety measurement method.

A portable finger pulse oximeter (Nellcor™ PMN10, Medtronic Corp. MN, USA) was used to measure the heart rate.

Data were statistically analyzed with the help of the Statistical Package for Social Sciences statistical software (SPSS 18.0), considering a 5% significance level. Nonparametric tests were used. Normality assumption was evaluated with the Kolmogorov Smirnov test. The association between two groups was analyzed by Wilcoxon Signed Rank Test.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 5-8 years
* Children who need at least two restorative dental treatments of the mandibular first primary molar

Exclusion Criteria:

* Chronic systemic illnesses
* Dental experience
* Mental disorders
* Invasive medical treatments
* Hospitalization
* Oral health problems with a painful history

Ages: 5 Years to 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: A total of 224 children aged 5-8 years who needed at least two restorative dental treatments of the mandibular first primary molar were included in the study. As the inclusion criteria, children with no mental disorders, with no past dental experience, hospitalization or invasive medical treatments, and no pain or symptom in their oral health. All included children and parents had to spoken and understood the Turkish language. Patients with chronic systemic illnesses that may affect the blood pressure or heart rate of a child were excluded from the study. Only children who required multiple-visit treatments were taken into consideration.
Sampling Method: Non-Probability Sample
Enrollment: 224 (Actual)
Dates: Start 2020-03-01 (Actual); Primary Completion 2020-07-30 (Actual); Study Completion 2020-08-30 (Actual)

PRIMARY OUTCOMES:
Dental anxiety | at the first dental visit, during two weeks
  The Modified Corah's Dental Anxiety Scale minimum 5 points maximum 25 points more than 15 points means patient have dental axiety .Higher points mean worse outcome
Dental anxiety | at the second dental visit, during two weeks
  The Modified Corah's Dental Anxiety Scale minimum 5 points maximum 25 points more than 15 points means patient have dental axiety .Higher points mean worse outcome

CONTACTS AND LOCATIONS:
Locations (1):
- Nurcan Kutluer Karaca, Erzincan, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No